CLINICAL TRIAL: NCT05529823
Title: The Effect of Showering During Labor on Perceived Labor Pain, Parenting Behavior and Birth Memory
Brief Title: Showering During Labor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sakarya University (Other)
Responsible Party: Principal Investigator, Yasemin Hamlaci Baskaya, Head of Midwifery Depatment, Sakarya University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 26082022
Record Dates: First submitted 2022-08-31; First posted 2022-09-07 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-07

CONDITIONS: Labor Pain; Parenting; Childbirth Problems
Keywords: Labor Pain; Birth Memories; Parenting Behavior; Hydrotherapy
MeSH Terms: conditions — Labor Pain

STUDY DESIGN:
Intervention Model Description: While warm showers will be used during labor in the experimental group, routine midwifery care will be applied in the control group.
Who Masked: Outcomes Assessor
Masking Description: Since there is no placebo group, masking only outcomes assessor.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The women in this group will have a warm shower during the labor process.
  Interventions: Behavioral: warm shower
- Control group (No Intervention): Women in the control group will not be interfered with and will be followed in line with the routine follow-up protocol of the clinic.

INTERVENTIONS:
Behavioral: warm shower — A warm shower will be applied for 20 minutes to the pregnant woman whose cervical dilatation reaches 4-5 cm and 7-8 cm.
  Arms: Experimental group

SUMMARY:
The research covers the birth memory evaluation to determine the pregnancy process, the labor process and the changes in the perceived pain level during this process, the parenting behavior immediately after the birth and the process of the birth.

DETAILED DESCRIPTION:
The Effect of Showering During Labor on Perceived Birth Pain, Parenting Behavior and Birth Memory Labor is a natural process in which the fetus and its appendages, which are the product of pregnancy, are expelled from the uterus approximately 40 weeks after the last menstrual bleeding. Birth is a very meaningful and unique experience for the pregnant woman and her family. Although it results in a positive experience, they are faced with serious pain, discomfort and sensory situations that will force them in this process. This pain is a severe acute pain and differs from other types of pain due to the fact that it is a part of a natural process, experienced in a limited time and mother-infant relationship. In the literature, labor pain can be relieved by two methods: pharmacological (drugs) and non-pharmacological (non-drug methods). In the guide published by the World Health Organization (WHO) in 2018, non-pharmacological methods are recommended to be used as they are more reliable and less invasive. Non-pharmacological methods are generally simple, reliable for mother-baby health, easy to use, accessible, economical and do not require special training. The application of non-pharmacological methods can be safely applied by midwives independently, as it does not require a physician's request and has minimal side effects. The midwife, who decides with the pregnant woman the non-pharmacological method to be used in the management of labor pain, can apply this method with her own autonomy and ensure that the mother has a more comfortable birth process. Non-pharmacological methods include hot/warm bath, hydrotherapy, hot-cold application, movement, positions, breathing, relaxation exercises, acupuncture, TENS, yoga, massage, aromatherapy, music, hypnosis. These practices increase the comfort of the pregnant woman during the labor process, relieve the level of pain and provide a positive birth experience and positive progress in the mother-baby interaction. One of the non-pharmacological methods used to reduce labor pain is hydrotherapy/warm application. Although there is not enough evidence about the history of Hydrotherapy/Hot treatment, it was reported that the spa waters of Hippocrates had a therapeutic effect in the fifth century. The use of water in childbirth and labor started with Igor Charkovsky in Russia in 1970, and then it was spread in Europe under the leadership of Micheal Odent. Hot application causes vasodilation in peripheral blood vessels, oxygenation of the region, nutrition, removal of waste materials, and relaxation is experienced by reducing tension in the muscles. In addition, the feeling of pain decreases. As a result, fetal well-being increases. The positive outcome of the birth process as a result of a healthy and beautiful progress also affects the understanding of mother-infant interaction and parenting behavior in the postpartum period. Postnatal parenting behavior is the behavior of the mother showing that she is interested in the newborn baby, such as taking care of the newborn in the postpartum period, asking questions about it, smiling at the newborn baby or making sounds. It can be affected by various factors, the situations experienced during labor and the past experiences of himself/herself. In a randomized controlled study conducted by Tuncay (2016), it was determined that the postpartum parenting behavior scale average score of the pregnants in the experimental group who received hydrotherapy was higher, and in other words, the pregnants in the experimental group behaved more positively towards the newborns in the postpartum period (p=0.001). Birth also affects memory. A pregnant woman who has experienced a difficult and long labor in the past is more anxious and fearful. However, past experiences do not always have this effect on women. Positive experiences with pain lead to correct behavior and positive changes. The experience experienced with the birth of each child is different and has the potential to change a woman's life in every sense. In order to protect the psychological health of the woman in the postpartum period, it is expected that her memories of the birth will be positive in her mind and that she will feel positive emotions when she remembers her birth. However, some women experience birth as a traumatic event rather than a positive and happy event. Some may describe this process as negative, while others may see it as a normal process. In the literature review, it has been determined that there are not enough studies on birth memory in Turkey. As a result, it is stated in the studies that non-pharmacological methods such as warm shower application may be effective in the positive outcome of labor, ensuring mother-infant interaction, acquiring parenting behavior and positive recall of labor in the future. For this purpose, the study was planned to evaluate the effect of warm shower applied during labor on women's pain levels, postpartum parenting behavior and birth memory.

ELIGIBILITY:
Inclusion Criteria:

* Being able to communicate verbally
* Between 18 - 45 years old,
* Being Primiparous/Nulliparous,
* Term pregnancy (38-41 weeks of pregnancy),
* Being in the latent and active phase of labor (Cervical dilation 4-5 cm and 7-8 cm)
* Having a single fetus
* Fetus in vertex presentation,
* Low risk pregnancy and no complications (EMR, Placenta Previa, HT, DM etc.),
* No obstetric risk (diabetes, pre-eclampsia, premature birth threat, etc.)
* Not having had any surgery in the spinal region,
* Volunteer to participate in the research

Exclusion Criteria:

* Not being willing to participate in the study,
* Not being open to communication and cooperation,
* Presence of hearing-sight and mental problems that would prevent the research,
* Be younger than 18 years old, over 45 years old,
* Being multiparous
* Being outside 38-41 weeks of gestation
* Being in the transitional phase of birth,
* Not planning a vaginal birth,
* Decision of cesarean delivery during labor,
* Presence of any medical or obstetric risk factors (fetal distress, prolonged labor, etc.)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 81 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-07-04 (Actual)

PRIMARY OUTCOMES:
Perceived pain level | 6 hours
  When cervical dilation is 4-5 cm and 7-8 cm, perceived labor pain will be defined by the visual pain scale.
Birth Memories and Recall Questionnaire | 6 hours
  It will be determined how taking a shower during labor will affect the birth memory.

SECONDARY OUTCOMES:
Postpartum Parenting Behavior Scale | 1 hours
  It will be determined whether taking a shower during labor affects parenting behavior.

CONTACTS AND LOCATIONS:
Locations (1):
- Sakarya Training and Research Hospital, Sakarya, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The follow-up of the study data will be provided by both researchers.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will be kept by the researchers until the study is reported. After the study is published, it will contribute to the literature.

REFERENCES:
- [Result] Britton HL, Gronwaldt V, Britton JR. Maternal postpartum behaviors and mother-infant relationship during the first year of life. J Pediatr. 2001 Jun;138(6):905-9. doi: 10.1067/mpd.2001.113358. PMID 11391337
- [Result] Callister LC. Making meaning: women's birth narratives. J Obstet Gynecol Neonatal Nurs. 2004 Jul-Aug;33(4):508-18. doi: 10.1177/0884217504266898. PMID 15346676
- [Result] Shaw-Battista J. Systematic Review of Hydrotherapy Research: Does a Warm Bath in Labor Promote Normal Physiologic Childbirth? J Perinat Neonatal Nurs. 2017 Oct/Dec;31(4):303-316. doi: 10.1097/JPN.0000000000000260. PMID 28520654
- [Result] Cluett ER, Burns E, Cuthbert A. Immersion in water during labour and birth. Cochrane Database Syst Rev. 2018 May 16;5(5):CD000111. doi: 10.1002/14651858.CD000111.pub4. PMID 29768662
- [Result] WHO recommendations: Intrapartum care for a positive childbirth experience. Geneva: World Health Organization; 2018. Available from http://www.ncbi.nlm.nih.gov/books/NBK513809/ PMID 30070803
- [Derived] Kulac V, Baskaya YH. The Effect of Showering During Labour on Perceived Labour Pain, Parenting Behaviour and Birth Memory: A Randomised Controlled Clinical Trial. Int J Nurs Pract. 2025 Oct;31(5):e70055. doi: 10.1111/ijn.70055. PMID 40930159